CLINICAL TRIAL: NCT04198532
Title: Effects of Contrast Bath on Sympathetic Skin Response in Patients With Complex Regional Pain Syndrome Type 1
Brief Title: Contrast Bath and Sympathetic Skin Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IstPMRTRHCRPSCB
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Stroke; Sympathetic Disorder
MeSH Terms: conditions — Stroke; Autonomic Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Regional Pain Syndrome(CRPS) group (Experimental): Stroke patients with complex regional pain syndrome
  Interventions: Other: Contrast bath
- Control Group (Other): Stroke patients without complex regional pain syndrome
  Interventions: Other: Contrast bath

INTERVENTIONS:
Other: Contrast bath — Contrast bath (hot and cold therapy)

SUMMARY:
This study evaluates the effects of contrast bath on sympathetic skin response in stroke patients with complex regional pain syndrome .

DETAILED DESCRIPTION:
Contrast bath(CB) is a thermal modality. It is usually performed by keeping hands in hot and cold water for certain periods of time. CB is a mostly advised intervention in complex regional pain syndrome (CRPS) altough there is no certain evidence The investigators will study on stroke patients. Change in sympathetic skin response after the contrast bath will be evaluated.

Stroke patients who admitted to the inpatient rehabilitation programme in Istanbul Physical Medicine and Rehabilitation Training and Research Hospital were evaluated for this study. Patients who had CRPS after stroke were included in the study (CRPS group). Also patients who had not CRPS and had similar age, gender and stroke duration with CRPS group were included in control group. Stroke patients with pacemaker, polyneuropathy, neglect, sensory or motor aphasia, peripheral nerve injury, hand surgery and reynauld disease were excluded from the study.

Age, gender, dominant arm, comorbidities, stroke side, aetiology and duration were recorded. Brunnstrom stages were used to evaluate arm and hand. Spasticity of upper extremity was assed by modified aschworth scale.

In CRPS group, CRPS severity scale was performed to evaluate the CRPS severity. This scale includes sensorial, autonomic and motor function. Also, neuropathic pain was assesed by Douleur Neuropathique 4 (DN4) Questionnaire and visual analog scale(VAS).

Contrast bath was performed to patients' plegic side . There were two baths , one include hot water and other had cold degrees. Patients hold their plegic hands in hot water for 4 minutes, in cold water for 1 minute after hot water. Hot and cold bath were repeated four times.

Sympathetic skin response (SSR) was measured before the contrast bath and 30 minutes after the contrast bath finished. SSR was recorded from plegic side and contralateral side. The active electrode was placed at the palm of the hand and the reference electrode at dorsum of the hand to record the median nerve SSR. The latency and the amplitude of SSR was measured.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* both gender

Exclusion Criteria:

* peripheral neuropathy
* pace maker
* skin lesion in hands
* anxiety
* sensory or motor aphasia
* peripheral nerve injury
* hand surgery and
* reynauld disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
sympathetic skin response | 1 day
  microvolts

CONTACTS AND LOCATIONS:
Overall Officials: Betul Yavuz Keles, MD, Study Director — Istanbul PMR training and research hospital; Burcu Onder, Assoc prof, Principal Investigator — Istanbul PMR training and research hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Physical Medicine and Rehabilitation Training and research Hospital, Istanbul
  - Istanbul PMR Training and Research Hospital, Istanbul

REFERENCES:
- [Derived] Yavuz Keles B, Onder B, Kesiktas FN, Ones K, Paker N. Acute effects of contrast bath on sympathetic skin response in patients with poststroke complex regional pain syndrome. Somatosens Mot Res. 2020 Dec;37(4):320-325. doi: 10.1080/08990220.2020.1830756. Epub 2020 Oct 14. PMID 33135537